CLINICAL TRIAL: NCT01697085
Title: Effects of Sea Buckthorn Oil on Mucous Membranes
Acronym: SBMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aromtech Ltd. (Industry)
Collaborators: The Finnish Funding Agency for Technology and Innovation (Unknown)
Responsible Party: Principal Investigator, Petra Larmo, R&D manager, Ph.D., Aromtech Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SBMM
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Mucous Membranes
Keywords: sea buckthorn; mucous membrane; dryness; metabolic syndrome; vaginal atrophy
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sea buckthorn oil (Experimental): 3 g (6 capsules)/day for three months
  Interventions: Dietary Supplement: Sea buckthorn oil
- Placebo oil (Placebo Comparator): 3 g (6 capsules)/day for three months
  Interventions: Dietary Supplement: Placebo oil

INTERVENTIONS:
Dietary Supplement: Sea buckthorn oil
  Arms: Sea buckthorn oil
Dietary Supplement: Placebo oil
  Arms: Placebo oil

SUMMARY:
Aim of this study is to investigate the effects of intake of sea buckthorn oil on mucous membranes

ELIGIBILITY:
Inclusion Criteria:

* women experiencing vaginal dryness
* 55-75 years of age
* at least 12 months from menstruation

Exclusion Criteria:

* use of estrogen replacement therapy

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in dryness related symptoms of genital mucous membranes | Interviews at baseline, at 2 months, at 3 moths (end of intervention), and daily during the study (symptom logbooks)
  Interview for symptom score at baseline and study visits and a daily symptom logbook during the intervention

SECONDARY OUTCOMES:
Change from baseline in vaginal pH | At baseline, at 3 months (end of intervention)

OTHER OUTCOMES:
Change from baseline in vaginal health index, vaginal dryness, vaginal maturity index, symptoms of dryness in other mucous membranes, markers of inflammation, oxidative stress and metabolic disorder in the circulation | At baseline, at 3 months (end of intervention)
  * Vaginal health index: index score, change from baseline
  * Vaginal dryness: moistening of pH test strip, change from baseline
  * Vaginal maturity index: change from baseline
  * Symptoms of dryness in other mucous membranes: daily symptom logbook during the intervention
  * Markers of inflammation, oxidative stress and metabolic disorders: analysis from serum/plasma, change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Risto Erkkola, Professor, Principal Investigator — Turun Gynekologikeskus, Turku, Finland
Locations (1):
- Turun Gynekologikeskus, Turku, Finland

REFERENCES:
- Available data/document: Clinical Study Report — http://www.maturitas.org/article/S0378-5122%2814%2900239-4/abstract?cc=y=